CLINICAL TRIAL: NCT00348673
Title: A Randomised, Double Blind, Placebo-controlled, Multicenter Study in Asymptomatic HIV Infected Patients to Investigate Pharmacodynamics, Pharmacokinetics, Safety and Toleration of UK-453,061
Brief Title: A Study in Asymptomatic HIV Infected Patients to Investigate Pharmacodynamics, Pharmacokinetics, Safety and Toleration of UK-453,061
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: A5271010
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-08

CONDITIONS: HIV-1
MeSH Terms: interventions — UK 453,061

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stage 1 (Experimental)
  Interventions: Drug: UK-453,061
- Stage 2 (Experimental)
  Interventions: Drug: UK-453,061

INTERVENTIONS:
Drug: UK-453,061 — Placebo BID, Placebo QD, UK-453,061 10 mg BID, 30 mg BID, 100 mg BID or 500 mg QD for 7 days
  Arms: Stage 1
Drug: UK-453,061 — Placebo BID, Placebo QD, UK-453,061 100 mg QD, 500 mg BID or 750 mg QD for 7 days
  Arms: Stage 2

SUMMARY:
A phase 2a study to investigate the effects of 7-day monotherapy of UK-453,061 on viral load response in asymptomatic human immunodeficiency virus (HIV) infected subjects, to assess the dose-response relationship, and to assess the pharmacokinetics (PK), safety and tolerability of UK-453,061 in asymptomatic HIV infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic HIV-1 infected male and patients aged 18-55 years inclusive.
* Patients with virus not containing NNRTI resistant mutations as determined by the VircoGEN virtual phenotyping essay.

Exclusion Criteria:

* Patients with a CD4 count less than 250 cells/mm3.
* Patients whose HIV infection has been diagnosed less than 3 months prior to screening, or for whom there is evidence of recent seroconversion.
* Patients with an HIV viral load less than 5000 copies/ml using RT-PCR(Roche Amplicor v1.5).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Germany (3):
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Hamburg

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271010&StudyName=A%20Study%20in%20Asymptomatic%20HIV%20Infected%20Patients%20to%20Investigate%20Pharmacodynamics%2C%20Pharmacokinetics%2C%20Safety%20and%20Toleration%20of%20UK-453%2C061%20

RESULTS

PARTICIPANT FLOW:
Groups:
- UK-453,061 10 mg Twice Daily (Stage 1): UK-453,061 10 milligram (mg) suspension orally twice daily for 7 days and as single morning dose on Day 8 in Stage 1.
- UK-453,061 30 mg Twice Daily (Stage 1): UK-453,061 30 mg suspension orally twice daily for 7 days and as single morning dose on Day 8 in Stage 1.
- UK-453,061 100 mg Twice Daily (Stage 1): UK-453,061 100 mg suspension orally twice daily for 7 days and as single morning dose on Day 8 in Stage 1.
- UK-453,061 500 mg Once Daily (Stage 1): UK-453,061 500 mg suspension orally once daily for 8 days in Stage 1.
- Placebo Once/Twice Daily (Stage 1): Placebo matched to UK-453,061 suspension orally once or twice daily for 7 days and as single morning dose on Day 8 in Stage 1.
- UK-453,061 750 mg Once Daily (Stage 2): Three UK-453,061 250 mg tablets, equivalent to 750 mg UK-453,061, along with 2 placebo tablets matched to UK-453,061 50 mg tablet orally once daily for 8 days in Stage 2.
- UK-453,061 500 mg Twice Daily (Stage 2): Two UK-453,061 250 mg tablets, equivalent to 500 mg UK-453,061, along with 1 placebo tablet matched to UK-453,061 250 mg tablet and 2 placebo tablets matched to UK-453,061 50 mg tablet orally twice daily for 7 days and as single morning dose on Day 8 in Stage 2.
- UK-453,061 100 mg Once Daily (Stage 2): Two UK-453,061 50 mg tablets, equivalent to 100 mg UK-453,061, along with 3 placebo tablets matched to UK-453,061 250 mg tablet orally once daily for 8 days in Stage 2.
- Placebo Once/Twice Daily (Stage 2): Three placebo tablets matched to UK-453,061 250 mg tablet along with 2 placebo tablets matched to UK-453,061 50 mg tablet orally once or twice daily for 7 days and as single morning dose on Day 8 in Stage 2.
Period: Stage 1
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | Placebo Once/Twice Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2) | Placebo Once/Twice Daily (Stage 2)
Started | 6 | 6 | 7 | 6 | 4 | 0 | 0 | 0 | 0
Treated | 6 | 6 | 6 | 6 | 4 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not Treated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | Placebo Once/Twice Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2) | Placebo Once/Twice Daily (Stage 2)
Started | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo matched to UK-453,061 suspension orally once or twice daily for 7 days and as single morning dose on Day 8 in Stage 1 or 3 placebo tablets matched to UK-453,061 250 mg tablet along with 2 placebo tablets matched to UK-453,061 50 mg tablet orally once or twice daily for 7 days and as single morning dose on Day 8 in Stage 2.
- Total: Total of all reporting groups
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2) | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (8.4) | 38.2 (8.6) | 33.5 (8.6) | 41.7 (4.1) | 29.2 (7.9) | 40.3 (7.5) | 37.0 (8.5) | 33.8 (8.0) | 36.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Human Immunodeficiency Virus-1 (HIV-1) Viral Load at Day 8
Description: Change from baseline in log 10-transformed plasma viral load(Human Immunodeficiency Virus-1 Ribonucleic Acid[HIV-1 RNA]) levels(log10 copies/milliliter[copies/mL])reported.Viral load determined using reverse transcriptase-polymerase chain reaction(RT-PCR) assay with standard lower limit of detection(LLOD) 400 copies/mL.For samples with reading less than (<)400 copies/mL,assay repeated using ultra sensitive method with LLOD of 50 copies/mL.Values below limit of quantification(LOQ) 50 copies/mL set to 50 copies/mL.Baseline was mean of three pre-dose values taken at screening,randomization,Day 1.
Time Frame: Baseline, Day 8
Population: Per protocol pharmacodynamic analysis set included all randomized participants who received at least 1 dose of study medication and had at least 1 post-dose viral load measurement.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
log10 copies/mL
  Baseline | 4.57 (0.33) | 4.39 (0.48) | 4.41 (0.27) | 4.38 (0.17) | 4.65 (0.46) | 4.55 (0.45) | 4.70 (0.33) | 4.57 (0.49)
  Change at Day 8 | -0.30 (0.20) | -0.78 (0.45) | -1.33 (0.38) | -1.67 (0.19) | -1.79 (0.32) | -1.62 (0.22) | -0.92 (0.38) | 0.01 (0.16)

2. Secondary Outcome: Number of Participants With Time to Rebound of Human Immunodeficiency Virus (HIV) Viral Load
Description: Time to rebound of viral load was defined as time from the last dose (Day 8) to the time of the first occasion at which the viral load was greater than baseline value. Number of participants with rebound of viral load at specified number of days after last dose (day 8) was reported.
Time Frame: Day 8 up to Follow-up (Day 38 to 40 [31 to 33 days post-last dose])
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants
  2 days | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  4 days | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  7 days | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  13 days | 1 | 2 | 4 | 3 | 3 | 1 | 0 | 0
  21 days | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
  31 to 33 days (follow-up) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1

3. Other Pre Specified Outcome: Area Under the Curve From Time Zero to End of Dosing Interval at Steady State (AUCtau,ss)
Description: AUCtau = Area under the plasma concentration versus time curve from time zero (pre-dose) to the end of the dosing interval (tau), the dosing interval was 12 hours for twice daily regimen and 24 hours for once daily regimen.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 12 hours post-dose; additional 24 hours post-dose for once daily regimen on Day 8
Population: Per protocol pharmacokinetic analysis set included all randomized participants who received at least 1 dose of study medication and had at least 1 post-dose pharmacokinetic concentration.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram*hour/milliliter (ng*hr/mL) | 47.2 (21.87) | 150.0 (51.57) | 686.7 (378.56) | 3543.5 (818.85) | 6530.1 (963.97) | 4719.4 (744.83) | 863.1 (260.83)

4. Other Pre Specified Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax,ss)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 12 hours post-dose; additional 24 hours post-dose for once daily regimen on Day 8
Population: as for outcome 3
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 14.6 (4.50) | 42.6 (20.31) | 146.6 (120.07) | 490.2 (248.68) | 1245.3 (560.17) | 979.1 (247.79) | 172.4 (51.53)

5. Other Pre Specified Outcome: Time to Reach Maximum Observed Plasma Concentration at Steady State (Tmax,ss)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 12 hours post-dose; additional 24 hours post-dose for once daily regimen on Day 8
Population: as for outcome 3
Measure: Median (Full Range); unit: hrs
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
hrs | 1.0 [1 to 3] | 1.0 [1 to 3] | 2.0 [1 to 4] | 3.0 [2 to 6] | 2.0 [1 to 3] | 1.5 [1 to 3] | 2.0 [1 to 3]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | UK-453,061 10 mg Twice Daily (Stage 1) | UK-453,061 30 mg Twice Daily (Stage 1) | UK-453,061 100 mg Twice Daily (Stage 1) | UK-453,061 500 mg Once Daily (Stage 1) | UK-453,061 750 mg Once Daily (Stage 2) | UK-453,061 500 mg Twice Daily (Stage 2) | UK-453,061 100 mg Once Daily (Stage 2) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 5/6 | 5/6 | 6/6 | 6/6 | 3/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UK-453,061 10 mg Twice Daily (Stage 1) (N=6) | UK-453,061 30 mg Twice Daily (Stage 1) (N=6) | UK-453,061 100 mg Twice Daily (Stage 1) (N=6) | UK-453,061 500 mg Once Daily (Stage 1) (N=6) | UK-453,061 750 mg Once Daily (Stage 2) (N=6) | UK-453,061 500 mg Twice Daily (Stage 2) (N=6) | UK-453,061 100 mg Once Daily (Stage 2) (N=6) | Placebo (N=6)
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UK-453,061 10 mg Twice Daily (Stage 1) (N=6) | UK-453,061 30 mg Twice Daily (Stage 1) (N=6) | UK-453,061 100 mg Twice Daily (Stage 1) (N=6) | UK-453,061 500 mg Once Daily (Stage 1) (N=6) | UK-453,061 750 mg Once Daily (Stage 2) (N=6) | UK-453,061 500 mg Twice Daily (Stage 2) (N=6) | UK-453,061 100 mg Once Daily (Stage 2) (N=6) | Placebo (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Chloropsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1
Feeling cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal chlamydia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anogenital warts (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Protein total increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 2 | 3 | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phlebolith (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.